CLINICAL TRIAL: NCT02027051
Title: Etude génétique Des Arméniens
Status: Completed | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C11-15; 2012-A00514-39 (Registry Identifier: IDRCB)
Record Dates: First submitted 2014-01-02; First posted 2014-01-03 (Estimated); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Healthy
Keywords: population genetics

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Saliva samples
Oversight: Data Monitoring Committee: No

SUMMARY:
This study aims at better understanding the genetic structure of the Armenians, an old population whose genetics has not been the subject of many studies. We will study 500 individuals whom grandparents originate from different regions of Armenia. Each individual will be genotyped using a large panel of genetic markers. Principal component analysis will be used to analyze the genetic structure of this population.

ELIGIBILITY:
Inclusion Criteria:

* Four grand-parents originating from Armenia

Exclusion Criteria:

* One or more grand-parents not originating from Armenia

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Descends of individuals originating from Armenia.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2014-06 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Genome wide genotyping of individuals | 3 months following inclusion

SECONDARY OUTCOMES:
Principal component analysis of genotypes | Three months after completion of individual genotypes

OTHER OUTCOMES:
Genetic structure | One month after principal component analysis of individuals

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuelle Genin, Researcher, Study Director — Institut National de la Santé Et de la Recherche Médicale, France
Locations (1):
- Hovnanian, Paris, France